CLINICAL TRIAL: NCT06992245
Title: Characterization of Placental Diffusion in Women With Diabetes Using DW-MRI
Brief Title: Characterization of Placental Diffusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0042-22-HYMC
Record Dates: First submitted 2022-12-05; First posted 2025-05-28 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy in Diabetic; Placenta Diseases
MeSH Terms: conditions — Pregnancy in Diabetics; Placenta Diseases | interventions — Diffusion Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: The 2 arms will include 3th trimester pregnant women. Group 1- diabetic pregnant women Group 2- low risk pregnant women
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregnant women with gestational diabetes mellitus (Experimental): 3Th trimester pregnant women with gestational diabetes mellitus
  Interventions: Diagnostic Test: DW-MRI
- Low risk pregnant women (Active Comparator): 3Th trimester pregnant women with unknown diseases (low risk factors)
  Interventions: Diagnostic Test: DW-MRI

INTERVENTIONS:
Diagnostic Test: DW-MRI — Predict changes in ovarian diffusion using DW-MRI scan

SUMMARY:
DW-MRI Allows a quantitative comparison of diffusion as an expression of tissue hypoxia. The investigators aim is to compare changes in placental diffusion in pregnant women with uncontrolled diabetes compared to healthy pregnant women using DW-MRI.

The investigators hypothesize that placentas of diabetic mothers will show lower diffusion / perfusion compared to placentas of healthy women.

DETAILED DESCRIPTION:
In highly uncontrolled diabetes there is an increased risk of intrauterine fetal death. The mechanism of fetal death is unknown and unpredictable. One of the theories points to hypoxia as a precursor to the death of the fetus in the womb. If the researchers succeed in predicting changes in the placenta with the help of MRI, it may be possible to understand the mechanism of fetal damage as well as in the future to develop a protocol for predicting pregnancies prone to fetal death in the womb.

ELIGIBILITY:
Inclusion Criteria:

* Women with PGAM (Pre-gestational diabetes) diagnosed before 20 weeks of pregnancy
* Women with GDMA (Gestational diabetes) diagnosed by OGTT after 20 weeks of pregnancy

Exclusion Criteria:

* pregnant women with placental hypoxia disease related in the past
* pregnant women with placental hypoxia disease related in the present
* non-singleton pregnancy
* women in active labor or rupture of membrane
* smoking women
* suspicion of placenta accreta

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 40 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Placental diffusion coefficient (D) measured by IVIM-DWI | Two years
  Placental diffusion coefficient (D, mm²/s) derived from intravoxel incoherent motion diffusion-weighted MRI (IVIM-DWI).
  Mean D values will be extracted from whole-placenta regions of interest and compared between parturients with poorly controlled diabetes and excessive fetal growth and low-risk parturients with appropriately grown fetuses.

SECONDARY OUTCOMES:
Placental perfusion fraction (f) measured by IVIM-DWI | Two years
  Placental perfusion fraction (f, unitless) derived from intravoxel incoherent motion diffusion-weighted MRI (IVIM-DWI).
  Mean f values will be extracted from whole-placenta regions of interest and compared between parturients with poorly controlled diabetes and excessive fetal growth and low-risk parturients with appropriately grown fetuses

CONTACTS AND LOCATIONS:
Overall Officials: Rinat Gabbay-Benziv, Prof, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hille Yaffe Medical Center, Hadera, Israel